CLINICAL TRIAL: NCT01242657
Title: Quit and Fit: Exploring the Effects of Physical Activity on Teen Smoking Cessation
Brief Title: Quit and Fit: Teen Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDCU48/CCU310821
Record Dates: First submitted 2010-11-11; First posted 2010-11-17 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco Use Cessation; Youth Tobacco Use; Physical Activity; Smoking Cessation Intervention
MeSH Terms: conditions — Tobacco Use Cessation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief Advice (No Intervention): Standard of care arm with no intervention; includes standard communication regarding youth tobacco cessation such as a brief discussion and printed materials
- Not On Tobacco (N-O-T) Program (Active Comparator): Teens randomized to this arm participated in the N-O-T program, a proven teen cessation program.
  Interventions: Behavioral: Not On Tobacco (N-O-T) Program
- Quit & Fit (Experimental): Teens randomized to this arm participated in the Not On Tobacco (N-O-T) program with an added physical activity module.
  Interventions: Behavioral: Physical Activity Module; Behavioral: Not On Tobacco (N-O-T) Program

INTERVENTIONS:
Behavioral: Physical Activity Module — Participants were provided pedometers in order to track specific "Step Goals", which were defined for male or female participants. In addition, each participant recorded other forms of physical activity in a "Challenge Log".
  Arms: Quit & Fit
Behavioral: Not On Tobacco (N-O-T) Program — Not On Tobacco (N-O-T) Program, a proven teen smoking cessation program
  Arms: Not On Tobacco (N-O-T) Program; Quit & Fit

SUMMARY:
The long term goal of the study entitled "Quit & Fit" was to revise, evaluate, and disseminate the American Lung Association´s (ALA) teen smoking cessation program called Not On Tobacco (N-O-T), with an added physical activity module. The physical activity module was intended to encourage youth to adopt a more physically active lifestyle. Research showed that physical activity may increase the odds of smoking cessation. The general N-O-T program goals are to help adolescents quit smoking; reduce cigarette use (for participants who are unable to completely quit); increase healthy lifestyle behaviors; and improve life skills such as stress management, decision making, communication, and interpersonal skills. The primary aim of the current research project was to reduce smoking among West Virginia teens. A two-prong secondary aim was to (a) increase participants´ physical activity behavior by supplementing the intervention with a physical activity component and (b) assess the mediating/moderating impact of physical activity on cessation outcomes. If participants quit smoking, the likelihood that they will develop smoking-related diseases is diminished. Participating in this project may aid smoking cessation and therefore improve participants´ health. Research was conducted among 19 of the 123 West Virginia public high schools. 236 teens were recruited to participate in the study over 3 years. This study is a clinical behavioral trial using a 3-group design, with subsequent random assignment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible to participate in this study if they:

  1. Volunteer to participate
  2. Are between the ages of 14-18
  3. Obtain written parental consent•
  4. Provide written assent
  5. Report smoking on at least 1 day in the past 30 days
  6. Speak and understand English •NOTE: Teens ages 18 or older will provide consent rather than assent. Parental consent will not be required.

Exclusion Criteria:

* WV high schools will be excluded from participating in the research study if school enrollment does not meet or exceed 300 students in grades 9-12.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 236 (Actual)
Dates: Start 2006-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Smoking cessation: quit and reduction rates | 6 months
  The primary aim of the current research project is to reduce smoking among West Virginia teens.

SECONDARY OUTCOMES:
Participants´ physical activity behavior | 6 months
  Increase participants´ physical activity behavior by supplementing the intervention with a physical activity component.
Impact of physical activity on cessation outcomes | 6 months
  Assess the mediating/moderating impact of physical activity on cessation outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Horn, EdD, Principal Investigator — West Virginia University; Melissa Taylor, MA, Study Director — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dino G, Horn K, Goldcamp J, Fernandes A, Kalsekar I, Massey C. A 2-year efficacy study of Not On Tobacco in Florida: an overview of program successes in changing teen smoking behavior. Prev Med. 2001 Dec;33(6):600-5. doi: 10.1006/pmed.2001.0932. PMID 11716656
- [Background] Dino G, Horn K, Abdulkadri A, Kalsekar I, Branstetter S. Cost-effectiveness analysis of the Not On Tobacco program for adolescent smoking cessation. Prev Sci. 2008 Mar;9(1):38-46. doi: 10.1007/s11121-008-0082-0. Epub 2008 Feb 20. PMID 18286372
- [Background] Branstetter SA, Horn K, Dino G, Zhang J. Beyond quitting: predictors of teen smoking cessation, reduction and acceleration following a school-based intervention. Drug Alcohol Depend. 2009 Jan 1;99(1-3):160-8. doi: 10.1016/j.drugalcdep.2008.07.011. Epub 2008 Sep 19. PMID 18804924
- [Derived] Horn K, Branstetter S, Zhang J, Jarrett T, Tompkins NO, Anesetti-Rothermel A, Olfert M, Richards T, Dino G. Understanding physical activity outcomes as a function of teen smoking cessation. J Adolesc Health. 2013 Jul;53(1):125-31. doi: 10.1016/j.jadohealth.2013.01.019. Epub 2013 Apr 9. PMID 23578440